CLINICAL TRIAL: NCT04236115
Title: Does Articaine, Rather Than Prilocaine, Increase the Success Rate of Anaesthesia for Extraction of Maxillary Teeth
Brief Title: Comparison of Articaine and Prilocaine for Extraction of Maxillary Teeth
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taibah University (Other)
Responsible Party: Principal Investigator, Giath Gazal, Associate Professor, Taibah University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Taibah dental College
Record Dates: First submitted 2020-01-15; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Overcoming the Failure of Anaesthesia; Maxillary Teeth; Dental Extraction
Keywords: Carticaine; dental extraction; injections; prilocaine
MeSH Terms: interventions — Epinephrine; Felypressin

STUDY DESIGN:
Intervention Model Description: double blinded randomised trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Articaine 4% with 1:00.000 Adrenaline (Active Comparator): if the patient was in articaine group, buccal infiltration technique was applied by inserting a short needle at the height of buccal sulcus along the long axis of the subject tooth for extraction.
  Interventions: Drug: Articaine 4%; Drug: Adrenalin
- Prilocaine with 3% Felypressin (0.03 I.U. per ml) (Active Comparator): if the patient was in prelocaine group, buccal infiltration technique was applied by inserting a short needle at the height of buccal sulcus along the long axis of the subject tooth for extraction.
  Interventions: Drug: Prilocain 3%; Drug: Felypressin

INTERVENTIONS:
Drug: Articaine 4% — Articaine 4% is dental local anaesthetic agent
  Arms: Articaine 4% with 1:00.000 Adrenaline
Drug: Prilocain 3% — prilocaine is dental local anaesthetic agent
  Arms: Prilocaine with 3% Felypressin (0.03 I.U. per ml)
Drug: Adrenalin — adrenaline is a vasoconstrictor
  Arms: Articaine 4% with 1:00.000 Adrenaline
Drug: Felypressin — Felypressin is a vasoconstrictor
  Arms: Prilocaine with 3% Felypressin (0.03 I.U. per ml)

SUMMARY:
Ninety-five patients, aged between 16 and 70 years old, were included in this study. Patients were divided into two groups. Group one received Articaine 4% with 1:00.000 Adrenalines. Group two received Prilocaine with 3% Felypressin (0.03 I.U. per ml). Onset time of anaesthesia was objectively evaluated by using electronic pulp testing.

DETAILED DESCRIPTION:
85 patients in this study had successful local anaesthetic followed by extraction within the study duration time (10 minutes). However, there were six patients with failure anaesthesia (5 in prilocaine group and 1 in articaine group). By application Person's Chi-square test (x2), there were no significant differences in the number of the episodes of the anaesthetic success between articaine and prilocaine groups at time intervals (P-value = 0.5). T- test showed there have been no important variations within the mean onset time of anaesthesia for articaine and prilocaine buccal infiltrations (P-value =0.1).

ELIGIBILITY:
Inclusion Criteria:

* Patients have one or two upper teeth for extraction, subject tooth or its adjacent must be vital, healthy patient or patient with mild systemic diseases (class I or II according to American Society of Anesthesiology).

Exclusion Criteria:

* Patients excluded from this study if they have allergy to local anaesthetic agents or need surgical, or multiple teeth extraction.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Does articaine, rather than prilocaine, increase the success rate of anaesthesia for extraction of maxillary teeth | 6 months
  to compare the anaesthetic performances of 3% prilocaine (the safest local anaesthetic) with 4 % articaine (the local anaesthetic with fastest onset time of action) when used for maxillary teeth extraction

CONTACTS AND LOCATIONS:
Locations (1):
- Taibah University, Madinah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
it will be provided on demand
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Gazal G. Does articaine, rather than prilocaine, increase the success rate of anaesthesia for extraction of maxillary teeth. Saudi J Anaesth. 2020 Jul-Sep;14(3):297-301. doi: 10.4103/sja.SJA_94_20. Epub 2020 May 30. PMID 32934619